CLINICAL TRIAL: NCT03991806
Title: Association of Centre of Excellence Self-Administered Questionnaire (CESAM) Score and Frailty Levels With Incident Health Adverse Events in Older Community Dwellers: Results of the Canadian Longitudinal Study on Aging
Brief Title: Association of Centre of Excellence Self- Administered Questionnaire Score and Frailty Levels
Status: Active, not recruiting | Type: Observational
Sponsor: Jewish General Hospital (Other)
Responsible Party: Principal Investigator, Olivier Beauchet, MD, Professor of Geriatrics, Jewish General Hospital
Other Study IDs: 2020-1844
Record Dates: First submitted 2019-06-14; First posted 2019-06-19 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Frailty; Cognitive Decline; Injuries; Fall Injury
MeSH Terms: conditions — Frailty; Cognitive Dysfunction; Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Obsservational — The frailty and the health adverse events of older adults will be assessed by using a questionnaire called: Association of Centre of Excellence Self-Administered questionnaire (CESAM).

SUMMARY:
This study evaluates the frailty and the health adverse events in the population of the Canadian Longitudinal Study on Aging. It will be used the Centre of Excellence Self-Administered questionnaire (CESAM) which assesses frailty of older adults by providing a score and a of frailty in 4 levels.

DETAILED DESCRIPTION:
Age is broadly recognized to confer a risk for health adverse outcomes, but it is an insensitive and non-specific measure for use in individual decision-making. Frailty has been emerging to take its rightful place as a better measure for over past decades. Despite general consensus that the concept of frailty is clinically useful, the lack of agreement on its definition and the challenge of its measurement by front-line health providers mean that frailty remains only 'their apparent' to chronological age as a criterion to select older persons at risk.

ELIGIBILITY:
Inclusion Criteria:

* Being 65 years and over
* Being enrolled in the Canadian Longitudinal Study on Aging

Exclusion Criteria:

* Never being enrolled in the Canadian Longitudinal Study on Aging
* Undisclosed health adverse events

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: In this research study take part people that are enrolled in the Canadian Longitudinal Study on Aging. Moreover, they are community dwellers who are frequently exposed to different health adverse events.
Sampling Method: Non-Probability Sample
Enrollment: 30000 (Estimated)
Dates: Start 2020-05-31 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Dementia | around 18 months
  The algorithm is a three- step process involving administration of the neuropsychological battery to develop composite score in the three domains-memory, executive function, and psychomotor speed.
  The primary outcome of the study will be to determine the number of participants to whom the memory, the executive function, and the psychomotor speed are affected.

SECONDARY OUTCOMES:
Medication | around 18 months
  In the maintaining contact interview, one question will be asked of all participants in relation to prescription medication use in the preceding month. A second question asks about the frequency of prescription drug use during this month.
  The secondary outcome of the study will be to determine the number of the medication that the participant take during a period of time.

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Beauchet, MD, Principal Investigator — Jewish General Hospital
Locations (1):
- Jewish General Hospital, Montreal, Quebec, Canada